CLINICAL TRIAL: NCT03604718
Title: Observational Prospective Study to Assess the Safety and Effectiveness Profile of Beltavac® Polymerized With Alternaria Alternata
Brief Title: Study to Assess the Safety and Effectiveness of Beltavac® Polymerized With Alternaria Alternata
Status: Completed | Type: Observational
Sponsor: Probelte Pharma S.L.U. (Industry)
Responsible Party: Sponsor
Other Study IDs: PRO-POL-2017-01; PRO-BEL-2017-01 (Other: AEMPS)
Record Dates: First submitted 2018-07-19; First posted 2018-07-27 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Rhinoconjunctivitis With or Without Allergic Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Beltavac® Polymerized with Alternaria alternata — Adminstration of Beltavac® Polymerized with Alternaria alternata according to the routine clinical practice

SUMMARY:
Non-interventional Study to Assess the Safety and Effectiveness Profile of a SCIT Therapy With Beltavac® Polymerized With Alternaria alternata in allergic patients

DETAILED DESCRIPTION:
This prospective open multi-centre non-interventional study assess the safety and effectiveness profile of the subcutaneous allergen-specific immunotherapy with Beltavac® Polymerized in Alternaria alternata allergic patients (children and adults) in routine medical care.

Patients receive a rush schedule administration every month for a year. They attend at least 4 study visits to inform about the adverse reactions, the self reported symptoms and the medication intake.

ELIGIBILITY:
Inclusion Criteria:

* Patients of the age of 5 years and older suffering from a clinically relevant Alternaria alternata induced allergic rhinitis
* Positive skin testing or IgE determination to the relevant allergen

Exclusion Criteria:

Patients suffering from acute or chronic infections or inflammations Patients suffering from uncontrolled asthma Patients with a known autoimmune disease Patients with active malignant disease Patients requiring beta-blockers Patients having any contraindication for the use of adrenaline

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from the age of 5 on, who suffer from allergic rhinoconjunctivitis caused by Alternaria alternata
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2018-06-07 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
Numbers of treatment-related local and systemic reactions | 1 year
  Number of adverse reactions occurred during the treatment period and classified according to the WAO standard

SECONDARY OUTCOMES:
Rhinoconjuntivitis medication intake | 1 year
  Medication intake for allergy symptons control at baseline, 6 and 12 months
Visual analogue Scale Score | 1 year
  Psycometric scale that assesses the global allergic disease discomfort. It is a 10 cm line representing severity from 0:"no symptoms" to 10 "highest level of symptoms"
IgE and IgG4 specific quantification | 1 year
  IgE and IgG4 quantification in serum measured at baseline, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Inmaculada Buendía Jiménez, Study Director — Probelte Pharma
Locations (13):
- Spain (13):
  - Universitary Hospital of Vic, Vic, Barcelona
  - Medical Center Fedear, Barcelona, Catalonia
  - University Hospital of Torrejon, Torrejón de Ardoz, Madrid
  - University Hospital of Cartagena, Cartagena, Murcia
  - Clínica de Alergia Mar Jiménez Lara, Talavera de la Reina, Toledo
  - Allergo Centre, Barcelona
  - Medical Center Cenvi Medic, Barcelona
  - Alergomundo, Madrid
  - Clinica Torrelodones, Madrid
  - Ojeda Clinic, Madrid
  - University Hospital Virgen de la Arrixaca, Murcia
  - Reina Sofia Universitary Hospital, Murcia
  - Clinica Alergologica Dr Moral, Toledo